CLINICAL TRIAL: NCT00724204
Title: Functional Evaluation of a Follow on Formula Supplemented With Lactobacillus Salivarius CECT5713
Brief Title: Safety Assessment of Lactobacillus Salivarius CECT5713 in 6 Months Old Children
Acronym: P010
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puleva Biotech (Industry)
Collaborators: Hospital Clinico Universitario San Cecilio (Other)
Responsible Party: Federico Lara-Villoslada, Puelav Biotech
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Safety Salivarius
Record Dates: First submitted 2008-07-28; First posted 2008-07-29 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Infection
Keywords: probiotics; safety; fecal microbiota; infections
MeSH Terms: conditions — Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): Children that consumed a follow on formula without Lactobacillus salivarius CECT5713
  Interventions: Dietary Supplement: follow on formula without probiotics
- B (Active Comparator): Children that consumed a follow on formula with Lactobacillus salivarius CECT5713
  Interventions: Dietary Supplement: follow on formula with Lactobacillus salivarius CECT5713

INTERVENTIONS:
Dietary Supplement: follow on formula without probiotics — A follow on formula without probiotics
  Arms: A
Dietary Supplement: follow on formula with Lactobacillus salivarius CECT5713 — follow on formula with Lactobacillus salivarius CECT5713 in a dose of 2x10E8 cfu/day
  Arms: B

SUMMARY:
The aim of the trial is to evaluate safety of a follow on formula supplemented with Lactobacillus salivarius CECT5713. A randomized double blind placebo controlled trial was carried out. Eighty six months old children were recruited by the department of pediatrics of Hospital Univeristario San Cecilio. Children were divided in two groups that consumed a follow on formula supplemented or not with the probiotic strain during 6 months. Fecal samples were obtained at the recruitment, at 3 months and at the end of the trial. In addition revision by the pediatrician was performed once a month and possible adverse effects were recorded both by the pediatrician and by parents.

ELIGIBILITY:
Inclusion Criteria:

* Healthy six months old children

Exclusion Criteria:

* Lactose intolerance
* Cow's milk protein allergy
* Serious metabolic diseases
* Antibiotic treatment
* Serious gastrointestinal diseases

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2006-04; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Adverse reactions | 3 months and 6 months

SECONDARY OUTCOMES:
growth parameters (height, length, head circumference) | 3 months and 6 months
Fecal microbiota | 3 months and 6 months
Fecal short chain fatty acids | 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: José A Maldonado, PhD, MD, Principal Investigator — Department of Pediatrics. Hospital Universitario San Cecilio; Mónica Olivares, PhD, Study Chair — Department of Nutrition and Health. Puleva Biotech. Granada; Federico Lara-Villoslada, PhD, Study Director — Department of Nutrition and Helath. Puleva Biotech. Granada
Locations (1):
- Hospital Universitario San Cecilio, Granada, Granada, Spain

REFERENCES:
- [Derived] Maldonado J, Lara-Villoslada F, Sierra S, Sempere L, Gomez M, Rodriguez JM, Boza J, Xaus J, Olivares M. Safety and tolerance of the human milk probiotic strain Lactobacillus salivarius CECT5713 in 6-month-old children. Nutrition. 2010 Nov-Dec;26(11-12):1082-7. doi: 10.1016/j.nut.2009.08.023. Epub 2009 Dec 16. PMID 20018483